CLINICAL TRIAL: NCT05878834
Title: Efficacy and Safety of Beta-glucan Supplement in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Oh87/65
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease Patients
Keywords: chronic obstructive pulmonary; beta-glucan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucan supplement group (Experimental): Beta-glucan supplement capsule composes of beta-glucan 250 mg, broccoli 75 mg, quercetin 50 mg.
  Interventions: Dietary Supplement: Beta-glucan supplement group
- Placebo group (Placebo Comparator): Placebo capsule is empty capsule.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Beta-glucan supplement group — Take 1 capsule 1 time per day for 12 weeks.
  Arms: Beta-glucan supplement group
Dietary Supplement: Placebo group — Take 1 capsule 1 time per day for 12 weeks.
  Arms: Placebo group

SUMMARY:
The objectives of this study are to evaluate Efficacy and safety of beta-glucan supplement in chronic obstructive pulmonary disease patients.

DETAILED DESCRIPTION:
There are 72 patients in this study. They are randomly divided into 2 groups which are beta-glucan supplement group and placebo group. The supplement will be taken 1 capsule/day for 12 weeks. Forced expiratory volume in 1 second/Forced vital capacity, Modified Medical Research Council Dyspnea Score, Breathlessness, Cough, and Sputum Scale, 6 Minute Walk Test, Diffusing capacity for carbon monoxide, Tumor necrosis factor alpha, Interleukin-6, C-reactive protein, glutathione, aspartate transaminase, alanine transaminase, alkaline phosphatase, creatinine, and blood urea nitrogen are assessed before and after taking supplement 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Chronic Obstructive Pulmonary Disease with Forced expiratory volume in 1 second/Forced vital capacity after receiving bronchodilator medicine more than 70%
* No exacerbation and uncontrolled disease
* 10 pack-years smoking history 10 pack-years but stop smoking more than 1 years
* Willing to participate in this study

Exclusion Criteria:

* Respiratory infection in 4 weeks
* Lung cancer
* Liver disease or kidney disease
* Lung surgery history
* Take kung supplement in 2 weeks
* Take warfarin, clopidogrel, aspirin, or digoxin
* Allergic to beta-glucan, broccoli, or quercetin
* Cannot use Spirometry
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second/Forced vital capacity | 12 weeks
  Forced expiratory volume in 1 second/Forced vital capacity in % (high value means better pulmonary function)

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Score | 12 weeks
  Modified Medical Research Council Dyspnea Score shows in dyspnea score (score 0 to 4 means low dyspnea to high severity).
Breathlessness, Cough, and Sputum Scale | 12 weeks
  Breathlessness, Cough, and Sputum Scale shows in severity scale (scale 0 to 4 means no symptom to high severity)
6-minute walk test | 12 weeks
  6-minute walk test in walking distance in 6 minutes (meters) (high value means better performance)
Chronic obstructive pulmonary disease assessment test | 12 weeks
  Chronic obstructive pulmonary disease assessment test in scale 0 to 5 (high value means better quality of life)
Tumor necrosis factor alpha | 12 weeks
  Tumor necrosis factor alpha is a pro-inflammatory cytokine (picogram/ml) (high value means high risk of inflammation)
Interleukin-6 | 12 weeks
  Interleukin-6 is a biomarker of inflammation (picogram/ml) (high value means high risk of inflammation)
C-reactive protein | 12 weeks
  C-reactive protein refers to inflammation (mg/ml) (high value means high risk of inflammation)
Aspartate transaminase | 12 weeks
  Aspartate transaminase refers to liver function (U/L)
Alanine transaminase | 12 weeks
  Alanine transaminase refers to liver function (U/L)
Alkaline phosphatase | 12 weeks
  Alkaline phosphatase refers to liver function (U/L)
Creatinine | 12 weeks
  Creatinine refers to renal function (mg/dl)
Blood urea nitrogen | 12 weeks
  Blood urea nitrogen refers to renal function (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Professor, Principal Investigator — Chulalongkorn University